CLINICAL TRIAL: NCT06674603
Title: The Trajectory and Influencing Factors of Cognitive Level in ICU Delirium Patients After Transfer Out of the ICU: Prospective Cohort Study
Brief Title: The Trajectory and Influencing Factors of Cognitive Level in ICU Delirium Patients After Transfer Out of the ICU
Status: Enrolling by invitation | Type: Observational
Sponsor: Zunyi Medical College (Other)
Collaborators: Guizhou Nursing Vocational College (Unknown)
Responsible Party: Principal Investigator, Yang Xia, researcher, Zunyi Medical College
Other Study IDs: gzwkj2024-253
Record Dates: First submitted 2024-09-17; First posted 2024-11-05 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-09

CONDITIONS: Cognition Disorder; ICU; Delirium
Keywords: ICU; delirium; cognition
MeSH Terms: conditions — Cognition Disorders; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ICU delirium patients

SUMMARY:
Introduction：Delirium is a prevalent psychiatric disorder observed in the Intensive Care unit(ICU) hat; often aggravates patients; overall health status, extends the duration of mechanical ventilation, prolongs ICU stays, and causes persistent or long-term cognitive impairment. A plethora of studies have indicated that the frequency, duration, and severity of delirium during hospitalization are significant risk factors for cognitive impairment in patients following transfer from the ICU. However, existing research has predominantly focused on cross-sectional analyses without delving into the influencing factors among patient subgroups. Consequently, the aim of this study is to employ the Latent Growth Curve Model (LGCM) and the Latent Class Growth Model (LCGM) model to analyze the trajectory of cognitive development and influencing factors of patients with delirium in the ICU one year after discharge.

Methods and analysis：This prospective study aims to investigate the trajectory of cognitive level variations of patients with delirium in ICU for one year. It is planned to recruit 240 participants and gather comprehensive data including general demographics, disease-related information, scores from the Minimum Mental State Examination, Hospital Anxiety and Depression Scale, and the Pittsburgh Sleep Quality Index. All data will be followed up using the same schedule on the day of transfer, 1 month after transfer, 3 months after transfer, 6 months after transfer and 1 year after transfer. Ultimately, the investigators will employ Latent Growth Curve Model and Latent Class Growth Model to analyze the trajectory of cognitive changes and identify potential categories, in addition to utilizing logistic regression modeling to explore influencing factors. The results of this study provide a theoretical framework for the clinical implementation of precision nursing interventions within this demographic, so as to prevent and reduce the decline of cognitive function and improve the quality of life of patients.

DETAILED DESCRIPTION:
A prospective longitudinal cohort study will be conducted in the ICU of a tertiary grade-A hospital in Guizhou Province. The study aims to recruit 240 patients diagnosed with ICU delirium, who were carefully selected based on predefined inclusion and exclusion criteria (Inclusion and exclusion criteria were as follows). The study is anticipated to commence in September 2024 and conclude in May 2026.

The inclusion criteria are:

1. Patients diagnosed with delirium by Confusion Assessment Model for Intensive Care Unit.
2. Age ≥ 18 years old.
3. Length of stay in ICU ≥24h.
4. Patients were able to complete the questionnaire by themselves or with the cooperation of their family members.5. Patients or family members gave informed consent and participated in the survey voluntarily.

The exclusion criteria are:

1. Previously diagnosed with dementia.
2. Mental illness or history of mental illness.
3. Suffering from traumatic brain injury, cerebrovascular disease, stroke, cranial surgery, intracranial infections, and other conditions that may affect cognitive function.
4. Presence of visual, hearing or communication impairments. Collection of general and disease-related information: trained staff assess ICU patients for delirium at the conclusion of the daily shift. Patients with delirium are included in the study, with the severity of delirium evaluated using the confusion assessment method for the ICU-7 scale. The date and time of delirium will be recorded, and the assessment will be carried out on a daily basis until the patient is transferred out of the ICU. Delirium-related information will be compiled after the patient's transfer out, and clinical subphenotypes of delirium will be ascertained using the RASS score , precipitant subphenotypes of delirium based on the patient's symptoms, severity of delirium based on the confusion assessment method for the ICU-7 scale, and the duration and frequency of occurrence of delirium based on the date and time of the recorded tracing. In addition, written informed consent will be obtained from the participants or their families prior to the commencement of data collection.

Follow-up data collection: at the time of patient transfer, the research team remains in contact with the participants and tracks their whereabouts and rehabilitation outcomes after discharge. Follow-up visits are conducted on the day of transfer (T1), 1 month after transfer (T2), 3 months after transfer (T3), 6 months after transfer (T4), and 1 year after transfer (T5) (see Table 4). Members of our study team will provide one-on-one contact with patients via WeChat video or face-to-face follow-up. Participants or family members are deemed disengaged if they are unwilling to cooperate in the study.

Outcome measures: cognitive level, anxiety and depression level and sleep status of delirium patients after discharge. Minimum Mental State Examination, Hospital Anxiety and Depression Scale and Pittsburgh sleep quality index will be used for measurement.

ELIGIBILITY:
The inclusion criteria are:

1. Patients diagnosed with delirium by CAM-ICU.
2. Age ≥ 18 years old.
3. Length of stay in ICU ≥24h.
4. Patients were able to complete the questionnaire by themselves or with the cooperation of their family members.
5. Patients or family members gave informed consent and participated in the survey voluntarily.

The exclusion criteria are:

1. Previously diagnosed with dementia.
2. Mental illness or history of mental illness.
3. Suffering from traumatic brain injury, cerebrovascular disease, stroke, cranial surgery, intracranial infections, and other conditions that may affect cognitive function.
4. Presence of visual, hearing or communication impairments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
cognitive level MMSE scale | from the day the patient was transferred out of the ICU to the end of the year.
  cognitive level will be assessed using the MMSE scale. The scale is designed to assess five aspects, namely orientation, memory, attention and calculation, recall, and language, with a total of score 30 points. The cognitive functioning improves as the score increases, with scores ranging from 27 to 30 being normal, and scores below 27 indicating cognitive dysfunction.The higher the score, the better the cognitive status of patients.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | from the day the patient was transferred out of the ICU to the end of the year.
  The scale is utilized for evaluating the extent of anxiety and depression present in patients.The scale contains 14 entries, including 2 subscales for anxiety and depression, with 7 entries rating depression and 7 entries rating anxiety. The total score of both subscales ranges from 0 to 7 for no anxiety or depression, 8 to 10 for critical anxiety or depression, and 11 to 21 for significant anxiety or depression.
Pittsburgh sleep quality index | from the day the patient was transferred out of the ICU to the end of the year.
  The scale evaluate a patient's quality of sleep in the last month. Each entry was rated on a scale of 0 to 3, summing up to a total score between 0 and 21, where higher scores signify a deterioration in sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Guizhou Vocational Nursing Technology College, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang X, Jiang Z, Chen F, Zhang X, Yuan X, Yang Y, Xu N, Li S. Trajectory and risk factors of cognitive level in ICU delirium patients after transfer out of the ICU: a protocol for a prospective cohort study. BMJ Open. 2025 Aug 12;15(8):e094232. doi: 10.1136/bmjopen-2024-094232. PMID 40803734